CLINICAL TRIAL: NCT01033708
Title: A Randomized Control Trial of Narrative Exposure Therapy Versus Treatment as Usual in the Therapy of Borderline Personality Disorder
Acronym: NET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zentrum für Integrative Psychiatrie (Other)
Collaborators: University of Konstanz (Other)
Responsible Party: Zentrum für Integrative Psychiatrie, Zentrum für Integrative Psychiatrie
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NET
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-10

CONDITIONS: Posttraumatic Stress Disorders; Borderline Personality Disorders
Keywords: Psychotherapy; PTSD; Borderline personality disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment as usual (Active Comparator): Treatment as usual
  Interventions: Behavioral: narrative exposure therapy
- narrative exposure therapy (Experimental): Narrative Exposure Therapy (NET), an evidence-based trauma-focussed treatment, suitable for survivors of prolonged and repeated exposure to traumatic stress and childhood adversities
  Interventions: Behavioral: narrative exposure therapy

INTERVENTIONS:
Behavioral: narrative exposure therapy — Narrative Exposure Therapy (NET), an evidence-based trauma-focussed treatment, suitable for survivors of prolonged and repeated exposure to traumatic stress and childhood adversities

SUMMARY:
Definition of the efficacy of NET compared with "treatment as usual" in the treatment of patients with complex traumatic disease (borderline personality disorder (BPD) and posttraumatic stress disorder (PTSD)) as assessed by structured clinical interviews. Furthermore, to evaluate the sleep, cortisol level and epigenetic differences in the process of the specific therapy compared to treatment as usual.

DETAILED DESCRIPTION:
Experimental intervention:

Narrative Exposure Therapy (NET), an evidence-based trauma-focussed treatment, suitable for survivors of prolonged and repeated exposure to traumatic stress and childhood adversity.

Control intervention:

Treatment as usual.

Follow-up per patient:

3 follow-up assessments- 4 weeks, 6 months,12 months and 24 months after end of experimental/ control intervention

Duration of intervention per patient:

Both treatment types will be conducted for 10-14 sessions of 60-90 min in length.

Additionally 5 sleep laboratory investigations (1 pre- and 4 post- intervention (4 weeks, 6 months, 12 months, 24 months after treatment)) will be carried out. Additionally the cortisol level in the hair and epigenetic markers will be recorded. The estimated observation time is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV -TR Diagnosis axis II: borderline personality disorder; axis I: posttraumatic stress disorder
* stable medication
* age 18-45 years, gender female
* legal competence
* sufficient cognitive function
* sufficient knowledge of the German or English language

Exclusion Criteria:

Known severe internal, neurological, musculoskeletal, endocrinological or sleep disorders with organic origin (clinical examination during the screening visit, judged by the investigator)

* gravidity (positive ß-HCG test)
* continuing and not interruptible exposure to sexual or physical abuse
* acute suicidal tendency
* positive drug-screening in urine toxicology test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | 0 - 1 - 6 - 12 - 24 month

SECONDARY OUTCOMES:
Borderline symptom checklist 23 (BSL) | 0 - 1 - 6 - 12 - 24

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum Integrative Psychiatrie, Kiel, Germany

REFERENCES:
- [Derived] Weinhold SL, Goder R, Pabst A, Scharff AL, Schauer M, Baier PC, Aldenhoff J, Elbert T, Seeck-Hirschner M. Sleep recordings in individuals with borderline personality disorder before and after trauma therapy. J Neural Transm (Vienna). 2017 Feb;124(Suppl 1):99-107. doi: 10.1007/s00702-016-1536-3. Epub 2016 Mar 12. PMID 26970970